CLINICAL TRIAL: NCT03691441
Title: Comparative Effectiveness Trial of Transoral Head and Neck Surgery Followed by Adjuvant Radio(Chemo)Therapy Versus Primary Radiochemotherapy for Oropharyngeal Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Charite University, Berlin, Germany (Other); University Medical Center Gießen and Marburg GmbH (Unknown); University Hospital Ulm (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TopROC
Record Dates: First submitted 2018-03-02; First posted 2018-10-01 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Oropharyngeal Cancer
Keywords: locally advanced; transorally resectable
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Radiotherapy; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, two-arm, open label, multicenter, randomized, controlled comparative effectiveness study.
  The trial is based on an event-driven design: the final analysis will be performed when all events have been observed or the study was terminated at one of the interim analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resection/adjuvant radio(-chemo)therapy (Experimental): * Transoral surgical resection within 4 weeks after randomization
  * Neck dissection can be performed during resection of the primary tumor or within 4 weeks after randomization
  * 6-7 weeks standard risk-adapted adjuvant radio(-chemo)therapy 56-66 Gy (chemotherapy according to arm B if necessary), start within 6 weeks post-surgery
  Interventions: Procedure: Resection; Radiation: Radiotherapy; Drug: Chemotherapy
- Adjuvant radio(-chemo)therapy/salvage neck dissection (Active Comparator): * 6-7 weeks standard radiotherapy (IMRT-technique), start within 4 weeks after randomization
  * 70-72 Gy, SIB possible
  * Cisplatin 100 mg/m2 on days 1, 22, 43 or Cisplatin once weekly (30-40 mg/m2) on days 1, 8, 15, 22, 29, 36 or Mitomycin C 10 mg/m2 d1, 29 and 5-FU 600 mg/m2/day iv on days 1-5 or Cisplatin 20 mg/m² + 5-FU 600 mg/m²/day iv d 1-5 and 29-33
  * +/- Salvage neck dissection 12±2 weeks after treatment
  Interventions: Radiation: Radiotherapy; Drug: Chemotherapy; Procedure: Salvage neck dissection

INTERVENTIONS:
Procedure: Resection — Definitive surgery should generally be performed within 2 weeks, but not more than 4 weeks after randomization. The appropriately indicated neck dissection(s) may be performed either prior to, during the same session, or within 2 weeks after the resection of the primary tumor, but not later than 4 weeks following randomization. The primary tumor is to be resected with clear margins (R0) and en bloc in all cases. Frozen section assessment must be routinely and readily available.
  Other Names: Transoral Surgery
  Arms: Resection/adjuvant radio(-chemo)therapy
Radiation: Radiotherapy — 6-7 weeks standard risk-adapted adjuvant radiotherapy 56-66 Gy, start within 6 weeks post-surgery Arm B: 6-7 weeks standard radiotherapy (IMRT-technique), start within 4 weeks after randomization, 70-72 Gy, SIB possible
Drug: Chemotherapy — The investigational medicinal product (IMP) are the chemotherapeutical drugs Cisplatin, Mitomycin C and 5-FU. According to local routine, chemotherapy protocols as listed in study protocol should be used.
Procedure: Salvage neck dissection — +/- Salvage neck dissection 12±2 weeks after treatment
  Arms: Adjuvant radio(-chemo)therapy/salvage neck dissection

SUMMARY:
Comparative Effectiveness Trial of Transoral Head and Neck Surgery followed by adjuvant Radio(chemo)therapy versus primary Radiochemotherapy for Oropharyngeal Cancer

DETAILED DESCRIPTION:
This trial investigates the effectiveness of transoral head and neck surgery (TOS) for locally advanced, but transorally resectable oropharyngeal cancer followed by risk-adapted adjuvant therapy versus primary radiochemotherapy (definitive chemoradiotherapy, CRTX). Both treatments are internationally accepted standards. The choice of the treatment strategy depends on the preference of the responsible attending physician and on the country of residence. Internationally, mostly definitive chemoradiotherapy is regarded as the standard of care for oropharyngeal cancer. In Germany, however, transoral surgical resection is also well established and commonly practiced. The key question therefore is whether one of the two therapies is more effective than the other in clinical daily routine under the given conditions of our health care system and with a realistic, non-ideal patient cohort. For this reason, a comparative effectiveness research (CER) concept will be applied in this setting. The aim of this trial is primarily to show a superiority of the surgical approach in terms of local and locoregional control and secondarily to compare functional outcome and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven SCC of the oropharynx; T1, N2a-c, M0; T2, N1-2c, M0; T3, N0-2c, M0, with only amendable to transoral resection)
* Primary tumor must be resectable through transoral approach
* p16 immunohistochemitry by local pathology or FFPE tissue must be available for central HPV diagnostic
* Written and signed informed consent
* Briefing through surgeon and radiation oncologist
* ECOG PS ≥2, Karnofsky PS ≥ 60 %
* Age ≥ 18
* Curative treatment intent
* Adequate bone marrow function: leucocytes > 3.0 x 109/L, neutrophils > 1.5 x 109/L, platelets > 80 x 109/L, hemoglobin > 9.5 g/dL
* Adequate liver function: Bilirubin < 2.0 g/dL, SGOT, SGPT, < 3 x ULN
* If of childbearing potential, willingness to use effective contraceptive method for the study duration and 2 months post-dosing.
* dental examination and appropriate dental therapy if needed prior to Confidential TopROC 2017_03_24 Version 1.0 Seite 15 von 124 beginning of radiotherapy
* Nutritional evaluation prior to initiation of therapy and optional prophylactic gastrostomy (PEG) tube placement

Exclusion Criteria:

* Prior invasive malignancy except controlled skin cancer or carcinoma in situ of cervix
* Unknown primary (CUP), nasopharynx, hypopharynx, laryngeal or salivary gland cancer
* Metastatic disease
* Serious co-morbidity, e.g. high-grade carotid artery stenosis, congestive heart failure NYHA grade 3 and 4, liver cirrhosis CHILD C
* Hemoglobin level <9.5g/dl within 4 weeks before randomization
* Pregnancy or lactation
* Women of child-bearing potential with unclear contraception
* Previous treatment with chemotherapy, radiotherapy, EGFR-targeting agents or surgery exceeding biopsy in head and neck
* Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days prior to study screening
* Social situations that limit compliance with study requirements or patients with an unstable condition (e.g., psychiatric disorder, a recent history of drug or alcohol abuse, interfering with study compliance, within 6 months prior to screening) or otherwise thought to be unreliable or incapable of complying with the requirements of the protocol
* Patients institutionalized by official means or court order
* Deficient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2024-05-05 (Estimated); Study Completion 2024-05-05 (Estimated)

PRIMARY OUTCOMES:
Time to local or locoregional failure or death from any cause | Defined as time from randomization up to 36 month
  The primary objective of this study is to evaluate the effectiveness of primary surgical versus non-surgical treatment of patients with locally advanced, but transorally resectable oropharyngeal cancer in terms of time to local or locoregional failure or death from any cause (LRF).

SECONDARY OUTCOMES:
Overall survival | Until 3 years after randomization
  Overall survival (OS) in both study arms, follow-up visits until the end of study
Disease-free survival | Until 3 years after randomization
  Disease-free survival (DFS) in both study arms. CT- Scans will be performed at month 3, month 6, 18, 30 and in case of suspicion of recurrence
Effectiveness in terms of toxicity | Until 3 years after randomization
  Effectiveness in terms of toxicity in both study arms. Monitoring of AE's/SAE's from randomization to 28 days after the last administration of IMP and/or 5 months after randomization in this trial
Effectiveness in terms of morbidity | Until 3 years after randomization
  Effectiveness in terms of morbidity (including swallowing function by MDADI Score) by late morbidity documentation in both study arms.
Quality of life evaluated by patient | Until 3 years after randomization
  Quality of life Questionnaires using QLQ H&N-43 in both study arms
Quality of life evaluated by patient | Until 3 years after randomization
  CareQuality of life Questionnaires using EORTC QLQ-C30 both study arms
Cost-utility | Until 3 years after randomization
  Cost-utility in both study armsusing Questionnaire Health Care Utilization and Productivity loss.
Cost-effectiveness | Until 3 years after randomization
  Cost-effectiveness in both study arms using Questionnaire Health Utilization and Productivity loss.

OTHER OUTCOMES:
Tertiary objectives include comparisons of treatment effects between HPV- Status | Up to 36 month
  Subgroup analysis of HPV-positive and HPV-negative oropharynx carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Jung Busch, PD Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (20):
- Germany (20):
  - Universitäts- HNO- Klinik Mannhein, Mannheim, Baden- Würtemberg
  - St. Vincentius- Kliniken Karlsruhe, Karlsruhe, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Helios Amper- Klinikum Dachau, Dachau, Bavaria
  - Ruppiner Klinken GmbH, Neuruppin, Brandenburg
  - Klinikum Ernst von Bergmann gemeinnützige GmbH, Potsdam, Brandenburg
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Gießen, Giessen, Hesse
  - Philipps-Universität Marburg, Marburg, Hesse
  - Elbekliniken Stade- Buxtehude GmbH, Klinikum Stade und Klinik Dr. Hancken, Stade, Lower Saxony
  - Klinikum Wolfsburg, Wolfsburg, Lower Saxony
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Kreiskliniken Gummersbach-Waldbröl GmbH Klinik Oberberg, Gummersbach, North Rhine-Westphalia
  - Katholischen Krankenhaus Koblenz, Koblenz, Rhineland-Palatinate
  - Universität des Saarlandes, Homburg, Saarland
  - Universitätsklinik Leipzig / Borna Sana Kliniken Leipziger Land, Leipzig, Saxony
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck, Schleswig-Holstein
  - Universitätsklinikum Jena, Jena, Thuringia
  - Berlin Charité, Berlin
  - Universitätsklinikum Hamburg Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehanna H, Beech T, Nicholson T, El-Hariry I, McConkey C, Paleri V, Roberts S. Prevalence of human papillomavirus in oropharyngeal and nonoropharyngeal head and neck cancer--systematic review and meta-analysis of trends by time and region. Head Neck. 2013 May;35(5):747-55. doi: 10.1002/hed.22015. Epub 2012 Jan 20. PMID 22267298
- [Background] Licitra L, Zigon G, Gatta G, Sanchez MJ, Berrino F; EUROCARE Working Group. Human papillomavirus in HNSCC: a European epidemiologic perspective. Hematol Oncol Clin North Am. 2008 Dec;22(6):1143-53, vii-viii. doi: 10.1016/j.hoc.2008.10.002. PMID 19010264
- [Background] Chaturvedi AK, Engels EA, Anderson WF, Gillison ML. Incidence trends for human papillomavirus-related and -unrelated oral squamous cell carcinomas in the United States. J Clin Oncol. 2008 Feb 1;26(4):612-9. doi: 10.1200/JCO.2007.14.1713. PMID 18235120
- [Background] Ang KK, Harris J, Wheeler R, Weber R, Rosenthal DI, Nguyen-Tan PF, Westra WH, Chung CH, Jordan RC, Lu C, Kim H, Axelrod R, Silverman CC, Redmond KP, Gillison ML. Human papillomavirus and survival of patients with oropharyngeal cancer. N Engl J Med. 2010 Jul 1;363(1):24-35. doi: 10.1056/NEJMoa0912217. Epub 2010 Jun 7. PMID 20530316
- [Background] Weinberger PM, Yu Z, Haffty BG, Kowalski D, Harigopal M, Brandsma J, Sasaki C, Joe J, Camp RL, Rimm DL, Psyrri A. Molecular classification identifies a subset of human papillomavirus--associated oropharyngeal cancers with favorable prognosis. J Clin Oncol. 2006 Feb 10;24(5):736-47. doi: 10.1200/JCO.2004.00.3335. Epub 2006 Jan 9. PMID 16401683
- [Background] Pfister DG, Spencer S, Brizel DM, Burtness B, Busse PM, Caudell JJ, Cmelak AJ, Colevas AD, Dunphy F, Eisele DW, Gilbert J, Gillison ML, Haddad RI, Haughey BH, Hicks WL Jr, Hitchcock YJ, Jimeno A, Kies MS, Lydiatt WM, Maghami E, Martins R, McCaffrey T, Mell LK, Mittal BB, Pinto HA, Ridge JA, Rodriguez CP, Samant S, Schuller DE, Shah JP, Weber RS, Wolf GT, Worden F, Yom SS, McMillian NR, Hughes M; National Comprehensive Cancer Network. Head and neck cancers, Version 2.2014. Clinical practice guidelines in oncology. J Natl Compr Canc Netw. 2014 Oct;12(10):1454-87. doi: 10.6004/jnccn.2014.0142. PMID 25313184
- [Background] Gregoire V, Lefebvre JL, Licitra L, Felip E; EHNS-ESMO-ESTRO Guidelines Working Group. Squamous cell carcinoma of the head and neck: EHNS-ESMO-ESTRO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2010 May;21 Suppl 5:v184-6. doi: 10.1093/annonc/mdq185. No abstract available. PMID 20555077
- [Background] Wegscheider K, Drabik A, Bleich C, Schulz H. [Benefit assessment in health services research and epidemiology]. Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz. 2015 Mar;58(3):298-307. doi: 10.1007/s00103-014-2106-1. German. PMID 25566839
- [Background] Lorincz BB, Mockelmann N, Busch CJ, Knecht R. Functional outcomes, feasibility, and safety of resection of transoral robotic surgery: single-institution series of 35 consecutive cases of transoral robotic surgery for oropharyngeal squamous cell carcinoma. Head Neck. 2015 Nov;37(11):1618-24. doi: 10.1002/hed.23809. Epub 2014 Aug 28. PMID 24955923
- [Background] Boscolo-Rizzo P, Gava A, Baggio V, Marchiori C, Stellin M, Fuson R, Lamon S, Da Mosto MC. Matched survival analysis in patients with locoregionally advanced resectable oropharyngeal carcinoma: platinum-based induction and concurrent chemoradiotherapy versus primary surgical resection. Int J Radiat Oncol Biol Phys. 2011 May 1;80(1):154-60. doi: 10.1016/j.ijrobp.2010.01.032. Epub 2010 Sep 23. PMID 20864267
- [Background] Hicks WL Jr, Kuriakose MA, Loree TR, Orner JB, Schwartz G, Mullins A, Donaldson C, Winston JM, Bakamjian VY. Surgery versus radiation therapy as single-modality treatment of tonsillar fossa carcinoma: the Roswell Park Cancer Institute experience (1971-1991). Laryngoscope. 1998 Jul;108(7):1014-9. doi: 10.1097/00005537-199807000-00012. PMID 9665249
- [Background] O'Hara J, MacKenzie K. Surgical versus non-surgical management of early stage oropharyngeal squamous cell carcinoma. Eur Arch Otorhinolaryngol. 2011 Mar;268(3):437-42. doi: 10.1007/s00405-010-1362-4. Epub 2010 Aug 27. PMID 20799040
- [Derived] Worthington HV, Bulsara VM, Glenny AM, Clarkson JE, Conway DI, Macluskey M. Interventions for the treatment of oral cavity and oropharyngeal cancers: surgical treatment. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD006205. doi: 10.1002/14651858.CD006205.pub5. PMID 37650478
- [Derived] Bussmann L, Laban S, Wittekindt C, Stromberger C, Tribius S, Mockelmann N, Bottcher A, Betz CS, Klussmann JP, Budach V, Muenscher A, Busch CJ. Comparative effectiveness trial of transoral head and neck surgery followed by adjuvant radio(chemo)therapy versus primary radiochemotherapy for oropharyngeal cancer (TopROC). BMC Cancer. 2020 Jul 29;20(1):701. doi: 10.1186/s12885-020-07127-2. PMID 32727416